CLINICAL TRIAL: NCT02515214
Title: Bariatric Surgery Registration in Women of Reproductive Age
Acronym: AURORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Roland Devlieger, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: AURORA
Record Dates: First submitted 2015-07-23; First posted 2015-08-04 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Bariatric Surgery Candidate; Pregnancy
Keywords: bariatric surgery; reproduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Breast milk samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of bariatric surgery has risen subsequently over the last decade, especially in women of reproductive age. (Unplanned) pregnancies in this subgroup are not rare because of e.g. an increased fertility (because of the weight loss) and a possible ineffectiveness of contraceptives (because of a malabsorption in the intestine). Although a pregnancy after bariatric surgery is generally known as safe, there are a few studies that indicate that a pregnancy after a bariatric surgery is not always without complications, and that it should be considered as a high risk pregnancy. The research on pregnancy outcomes after this type of surgery is rather limited to a few small, mainly retrospective, observational case-control and cohort studies and a limited amount of case studies. For risk- and prognose related issues, e.g. the effect of bariatric surgery on fertility, timing of the pregnancy, development of complications during the pregnancy and pregnancy outcomes, large prospective cohort studies are needed. Besides, breast feeding practices and breast milk composition have scarcely been investigated in this population. The energy content of breast milk could possibly be influenced by a state of malabsorption after the procedure. Low amounts of vitamin B12 have also been noticed in the breast milk of women the surgery. The overall objective of this study is to establish a group of women at reproductive age (age 18-45) with a history of bariatric surgery and to generate an extensive database for future analysis. The final goal of the researchers is to develop guidelines or recommendations on how to manage pregnancies after bariatric surgery, based on large-scale prospective research.

The study design is a multicentric observational and prospective cohort study. Participants will be followed from the moment of surgery until 6 months postpartum and they can be included on several time points (before surgery, after surgery (<12 months); after surgery (>12 months) or during the pregnancy). Both retrospective and prospective data concerning the medical background, fertility (menstrual cycle), lifestyle (e.a. food, physical activities, smoking, sleeping), blood samples, psychological factors (fear and depression), sexuality, quality of life and pregnancy outcomes will be collected. Data collection by the investigators will happen in a web-based database and by direct online registration by the subjects.

DETAILED DESCRIPTION:
The investigators aim to develop guidelines or recommendations for the management of pregnancies after bariatric surgery based on large-scale prospective research.

The investigators want to:

1. investigate pregnancy outcomes of women with a history of bariatric surgery according to procedure, interval between surgery and conception, weight change after surgery and during pregnancy and nutritional status, taking into account possible confounding factors such as economic status, alcohol and tobacco use, sleep duration, psychological factors (anxiety and depression) and quality of life
2. determine the incidence of nutritional deficiencies in (pregnant) women of reproductive age after bariatric surgery.
3. evaluate the effect of bariatric surgery in (morbidly) obese women of reproductive age on anthropometry, fertility, sexuality, co-morbidities, use of medication and contraceptives, pregnancy outcomes, quality of life, psychological factors (anxiety and depression), blood biochemical parameters (nutritional status), food intake and physical activity
4. examine breastfeeding practices (intention, initiation, duration) and breast milk composition in women with a history of bariatric surgery

The study is a multicentric prospective cohort study with UZ Leuven as the coordinating central cite and AZ St Jan Brugge (obesity clinic and obstetric clinic), AZ St Lucas Brugge (obstetric clinic), AZ St Nikolaas St Niklaas (obesity clinic), UZ Gent (obesity clinic and obstetric clinic), AZ St Augustinus Wilrijk (obstetric clinic) and CHRH Mons Hainaut (obesity clinic and obstetric clinic) as local sites.

The design for the breast milk analyses is longitudinal and will, for practical reasons, only be initiated in UZ Leuven and UZ Gent. The investogators will collect a breast milk sample of 10 ml on day four of the postpartum and then weekly by the participants at home until the routine 6 week postpartum consultation.

Women will be included in one of the following four inclusion moments (IM):

* Before surgery (women of reproductive age with morbid obesity) (IM1)
* After surgery and not being pregnant (IM2)
* Before 15 weeks of gestation (IM3)
* Day 3 of 4 of the postpartum for breast milk analyses (IM4)

A simple, user-friendly website will be used to simplify the collection and entry of data and to create a large database. Researchers will be able to directly and continuously register patient data (replacing paper forms) and participants will be able to complete the questionnaires online. The database will be available via a secure online login. Participating researchers will only have access to their own patient database.

For breast milk analyses, the investigators wil collect a sample of 10 ml during the first feeding moment (between 8 am and 11am) on day four of the postpartum manually or by use of a vacuum pump. Each sample is divided into two different recipients. One part of the sample is frozen immediately in the freezer at -20 °C. The rest of the sample will immediately be heated to +40 °C by use of a bottle warmer. As soon as the sample is heated, it will be ultrasonically analyzed with the MIRIS Sonicator® in order to ensure that the sample is homogeneous. Immediately afterwards, the sample is analyzed with the Human Milk Analyzer (HMA) (MIRIS ®, Uppsala, Sweden) for fat (g/100 ml), proteins (g/100 ml), carbohydrates (g/100 ml), dry matter (g/100 ml) and energy (kcal/100ml). The samples that are being collected at the participants' homes will be frozen at -20° and afterwards analyzed with the HMA.

There are eleven measurement points:

T0 = baseline T1 = pre-operative T2 = 3 weeks post-operative T3 = 3 months post-operative T4 = 6 months post-operative T5 = 12 of x months post-operative T6 = first trimester pregnancy T7 = second trimester pregnancy T8 = third trimester pregnancy T9 = pregnancy T10 = 6 weeks postpartum T11 = 6 months postpartum The number of measurements varies according to the moment of inclusion.

1. Demographical data will be collected at (T0) (participant self-reporting). Age, nationality, ethnicity, marital status, family status, educational level, employment status and profession wil be questioned.
2. Anthropometric data, including body weight, waist circumference, hip circumference and body fat percentage (if measured) are collected at all measurement points and will be recorded by the researcher. The body length is only questioned at the first measurement. Body height and body weight will be used to calculate the Body Mass Index (kg/m²) at each measurement point.
3. During the first measurement the investigators will ask for past medical conditions (reported by the researcher) and obstetric history (gravidity, parity, abortion - self-report participant);
4. The type of procedure, date of surgery and institute of the surgeon will be recorded by the investigators during the first measurement (Reported by researcher). Potential problems or complications will be reported at the next measurement points. (T1-T5).
5. Current medical conditions (eg hypertension) will be reported at each measurement point, together with the used medication (Reported by the researcher).
6. The nutritional status of the participant will be assessed by the investigators on the basis of biochemical parameters in the venous blood. The nutritional status of the newborn will be assessed on the basis of biochemical parameters in the venous umbilical cord blood.

   (total protein and albumin, fasten glucose level, fat soluble vitamins A, 25 -hydroxy- vitamin D, vitamin E and vitamin K1, water soluble vitamins B1, vitamin B12 and folate (in the serum and red blood cells (RBC), iron , (+ transferrin, transferrin saturation, ferritin ), calcium, zinc and magnesium, hematology (hemoglobin, hematocrit and RBC count, mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV)), coagulation (prothrombin time (PT) and activated partial thromboplastin time (aPTT)).

   During measurement time T1, T3, T4, T5, a blood sample will be taken at the department of endocrinology and on T6, T7, T9 and T10 at the department of obstetrics-gynecology.
7. Investigators will ask the participants about alcohol, tobacco and sleeping habits (self-report participant). The alcohol consumption will be asked by using the AUDIT-C questionnaire (Alcohol Abuse Disorder Identification Test). If the participant smokes, the amount of cigarettes or other tobacco products that are smoked daily will be recorded.

   At the beginning of pregnancy, the participant will be asked whether alcohol and tobacco use have changed. Finally, the sleep duration will also be determined.
8. The food intake will be measured during three days (of which at least 1 day in the weekend), on the basis of a 3-day food diary (self-report participant). The intake of supplements is also questioned (self-report participant).
9. Physical activity will be measured by use of the Kaiser Physical Activity Survey (KPAS), a modified version of the Baecke physical activity questionnaire, which was specifically designed to assess the physical activity in women. The KPAS assesses different domains of physical activity (household /family care activities, professional activities, activities of daily life and sports/exercise). The KPAS was validated for both pregnant and non-pregnant women.
10. The Moorehead-Ardelt Quality of Life Questionnaire II (MA QoLQII) will be used both pre-and postoperatively to assess the quality of life (self-report participant). This validated questionnaire is part of the Bariatric Analysis and Reporting Outcome System (BAROS). The MA QoLQII has been validated in an obese population and can be used for bariatric surgery.
11. The Self-Rating Questionnaire will be used to assess the psycho-social condition of the participant. This is a Dutch-validated questionnaire to measure anxiety, based on the American "State-Trait Anxiety Inventory" version Y of Spielberger (35). The questionnaire included two separated self- questionnaires in which two different concepts can be measured: state anxiety and trait anxiety. The Edinburgh Depression Scale (EDS), a validated 10-item questionnaire, will be used to measure depression during pregnancy and postpartum (self-report participant).
12. A questionnaire will be used to record the menstrual cycle (self-report participant). The menstrual cycle's length, duration of bleeding, number of periods per year, the pattern of the menstrual cycle and the presence of amenorrhea or oligomenorrhea will be assessed. The questionnaire is administered at T1, T4 and T5.
13. Pregnancy intention is asked in non-pregnant women (self-report participant) at the first measurement point (T0).
14. The use of contraceptives, which also examines the therapy adherence, is also questioned (self-report participant). The questionnaire is administered at T1, T4 and T5.
15. Sexuality will be questioned to determine the relationship with fertility and the interval between surgery and pregnancy (self-report participant). The questionnaire will be completed at T1, T4 and T5.
16. Clinical pregnancy outcomes of the mother will be questioned each pregnancy trimester (T6-T8) (Reported by the researcher) e.g. conception method, blood pressure, gestational age, gestational diabetes, pre-eclampsia, pregnancy-induced hypertension, clinical problems, etc. The results of the fetal ultrasounds will also be collected during each pregnancy trimester (T6-T8). During childbirth (T9) the duration of pregnancy, labor and delivery method will be questioned. The parameters of the newborn, including gender, birth weight, birth length, head circumference, Apgar scores, admission to the neonatal intensive care unit (NICU) and any complication will be recorded (T9). Finally, postpartum data such as hemoglobin, prescribed supplements, breastfeeding, or any other problems will be recorded.
17. A structured questionnaire about breastfeeding practices, developed by Guelinckx et al. (2011), will be used at 6 months postpartum (T11) (self-report participant). This questionnaire consists of 11 questions including the intention to breastfeed, breastfeeding initiation, duration of (exclusive) breastfeeding and the reasons to stop with breastfeeding.

ELIGIBILITY:
Women will be included in one of the following four inclusion moments (IM):

* Before surgery (women of reproductive age with morbid obesity) (IM1)
* After surgery and not being pregnant (IM2)
* Before 15 weeks of gestation (IM3)
* Day 3 of 4 of the postpartum for breast milk analyses (IM4)

Inclusion and exclusion criteria:

1. IM1

   Inclusion criteria:
   * Women
   * Age between 18 and 45 years
   * planning bariatric surgery

   Exclusion criteria:

   - Infertile (eg, hysterectomy, menopause, etc.)
2. IM2

   Inclusion criteria:
   * Women
   * Age between 18 and 45 years
   * A bariatric surgery in the past

   Exclusion criteria:

   - Infertile (eg, hysterectomy, menopause, etc.)
3. IM3

   Inclusion criteria:
   * Women
   * Age between 18 and 45 years
   * A bariatric surgery in the past
   * <15 weeks pregnant

   Exclusion criteria:

   - Recruitment after 15 weeks of gestation
4. IM4

Inclusion criteria:

* Women
* Age between 18 and 45 years
* A bariatric surgery in the past
* Gestational age between 37 and 42 weeks
* Giving birth of a viable child (singleton)
* Breastfeeding on day 3 of the postpartum

Exclusion criteria:

* Intake of the following drugs during lactation: psychotropic drugs, cytotoxic drugs, beta-blockers, dopamine agonists, aspirin, antihistamines, ergotamine, lithium, phenindione, barbiturates, anticonvulsants and sulfasalazine
* Diabetes mellitus or diabetes mellitus gravidarum
* Newborn admitted to the NICU (no rooming-in)
* Uncertainty if milk production is sufficient to meet the needs of the baby (in consultation with the midwife)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Women of reproductive age attending for bariatric surgery
  2. Women of reproductive age with a history of bariatric surgery
  3. Pregnant women with a history of bariatric surgery
  4. Lactating women with a history of bariatric surgery
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-07; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | Birth
  Weight at birth minus weight at start of pregnancy
Gestational length | Birth
  Preterm (<37w of gestation) vs a term (37-42w of gestation) delivery
Surgical complications during pregnancy | up to birth
  bowel obstruction, strangulation, internal herniation
Gestational diabetes mellitus | up to birth
  disturbed glucose metabolism
Hypertensive disorders | up to birth
  pregnancy-induced hypertension, (pre-)eclampsia
Birth weight | Birth
  Weight of newborn baby (<2.5kg small-for-gestational age; >4kg macrosomia)

SECONDARY OUTCOMES:
Quality of life assessed by the Moorehead-Ardelt Quality of Life Questinnaire II | preoperatively, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6w and 6 mo)
  quality of life assessed by the Moorehead-Ardelt Quality of Life Questinnaire II
Breast milk fat content | weekly from day 3-4 after delivery until week 6 after delivery
  Breast milk fat content assessed by the Human Milk Analyzer
Contraception | baseline, postoperatively (6 and 12mo)
  Pattern and duration of menstrual cycle and contraceptive use assessed by a self-developed questionnaire
Physical activity | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6 mo)
  Level of physical activity (household, work, free time, sports) assessed by the Kaiser Physical Activity Survey
Dietary intake | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6 mo)
  Dietary intake assessed by a semi-structured 3 day estimated dietary record method (3 day food diary)
Sleeping habits | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6 mo)
  sleeping habits (week and week-end) assessed by a self-developed questionnaire
Breastfeeding practices | Postpartum period (6mo)
  Assessed by a structured questionnaire by Guelinckx et al. (2011): initiation and duration of breastfeeding, exclusively breastfeeing, artificial feeding
Anxiety | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 3 (28-32w) and postpartum period (6w and 6 mo)
  State and Trait anxiety assessed by the State-Trait Anxiety Inventory
Depression | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 3 (28-32w) and postpartum period (6w and 6 mo)
  depressive feelings assessed by the Edinburgh Postnatal Depression Scale;
Alcohol use | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6 mo)
  drinking habits assessed by the Alcocol Abuse Disorder Identification Test (AUDIT-c)
Smoking habits | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w) and 3 (28-32w) and postpartum period (6 mo)
  Smoking habits (amount of sigarets, changes during pregnancy) assessed by a self-developed questionnaire
Sexuality | baseline, postoperatively (6 and 12mo)
  Sexual activity is assessed by a self-developed questionnaire
Total blood count | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  red blood cells, hematocrit, hemoglobin, MCV, MCH, MCHC assessed by venipuncture
Vitamin A | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Vitamin A serum level assessed by venipuncture
25-OH-vitamin D | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Vitamin 25-OH-vitamin D serum level assessed by venipuncture
vitamin K1 | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Vitamin K1 serum level assessed by venipuncture
Vitamin B-12 | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Vitamin B12 serum level assessed by venipuncture
Folate | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Folate (serum and red blood cells) assessed by venipuncture
Coagulation | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  prothrombin time, activated partial tromboplastin time and coagulation factors assessed by venipuncture
Glucose | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Fasten glucose level assessed by venipuncture
Zinc | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Zinc serum level assessed by venipuncture
Anemia | baseline, postoperatively (6 and 12mo), pregnancy trimester 1 (12w) and 2 (20-24w) and postpartum period (6w)
  Iron, ferritin, transferrin (saturation) levels assessed by venipuncture
Breast milk protein content | weekly from day 3-4 after delivery until week 6 after delivery
  Breast milk fat protein assessed by the Human Milk Analyzer
Breast milk carbohydrate content | weekly from day 3-4 after delivery until week 6 after delivery
  Breast milk carbohydrate content assessed by the Human Milk Analyzer
Breast milk energy content | weekly from day 3-4 after delivery until week 6 after delivery
  Breast milk energy content assessed by the Human Milk Analyzer
Mode of delivery | Birth
  vaginal, cesarean section, instrumental delivery
Apgar score | Birth (2-5-10 minutes)
  Apgar score (appearance, pulse, grimase response, activity, respiration) assessed by the medical staff
Body weight | baseline, post-operatively (3w, 3, 6 and 12mo), pregnancy trimester 1 (12w), 2 (20-24w), and 3 (28-32w) and the postpartum period (6w and 6mo)
  Weight measured by the medical staff to 1) calculate the body mass index and 2) to report weight loss (after surgery) or weight gain (during pregnancy)

OTHER OUTCOMES:
Maternal age | baseline
  Maternal age (birth date, age) assessed by online questionnaire
Nationality | baseline
  Belgium versus other assessed by online questionnaire
Family status | baseline
  Family status (living together with or without children, living seperate, living with parents) assessed by online questionnaire
Educational level | baseline
  Educational level (until 18 yr, +18yr high school, +18yr university or higher) assessed by online questionnaire
Profession | baseline
  Profession (working full/half time, studying, unemployed) assessed by online questionnaire
Marietal status | baseline
  Marietal status (married, living together, in a relation, divorced, widow) assessed by online questionnaire
BMI | baseline
  body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Roland Devlieger, MD, PhD, Principal Investigator — KU Leuven, Dpt. Of Development and Regeneration; UZ Leuven, Dpt. of Obstetrics and Gynecology
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Jans G, Devlieger R, De Preter V, Ameye L, Roelens K, Lannoo M, Van der Schueren B, Verhaeghe J, Matthys C. Bariatric Surgery Does Not Appear to Affect Women's Breast-Milk Composition. J Nutr. 2018 Jul 1;148(7):1096-1102. doi: 10.1093/jn/nxy085. PMID 29901782
- [Derived] Jans G, Matthys C, Bel S, Ameye L, Lannoo M, Van der Schueren B, Dillemans B, Lemmens L, Saey JP, van Nieuwenhove Y, Grandjean P, De Becker B, Logghe H, Coppens M, Roelens K, Loccufier A, Verhaeghe J, Devlieger R. AURORA: bariatric surgery registration in women of reproductive age - a multicenter prospective cohort study. BMC Pregnancy Childbirth. 2016 Jul 29;16(1):195. doi: 10.1186/s12884-016-0992-y. PMID 27473473
- See also: Communication platform AURORA study — http://www.aurorastudy.org/en